CLINICAL TRIAL: NCT04814992
Title: Pre-op CBT to Reduce the Risk for Development of Chronic Post-surgical Pain in Patients Undergoing Total Knee Arthroplasty
Brief Title: Pre-op Cognitive Behavior Therapy to Decrease Chronic Post-Surgical Pain in TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Peggy Compton, RN, PhD, Associate Professor, van Ameringen Endowed Chair, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 844378
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: Chronic Post-Surgical Pain
Keywords: CPSP; Chronic Post-Surgical Pain; Cognitive Behavioral Therapy; Total Knee Arthroplasty; Motivational Interviewing; Opioid Taper
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial is proposed to evaluate the efficacy of the novel computer-assisted preoperative CBT with integrating motivational interviewing intervention to affect acute and chronic post-operative pain outcomes. Specifically, 90 adult patients over the age of 21 meeting study inclusion criteria and preparing to undergo TKA at the Department of Orthopedic Surgery at Penn Presbyterian Medical Center, Penn Medicine University City, Penn Medicine Radnor, and Pennsylvania Hospital will be randomized to either receive the computer-assisted preoperative CBT intervention (n=45) or treatment-as-usual (control, n=45).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer-Assisted Preoperative CBT Intervention (Active Comparator): Patients will receive the computer-assisted preoperative CBT intervention (n=75). A particularly promising internet-based CBT pain program for the population of interest, PAINTrainer, demonstrated improved pain, function, coping and global health in patients with chronic knee arthritic pain in comparison to an internet education control, with benefits persisting for up to 52 weeks. In addition to the PAINTrainer, there will be an integration of a motivational interviewing (MI) intervention delivered by a trained "coach" across the sessions about (1) the benefits of opioid tapering for post-operative pain control, (2) approaches for safely tapering, (3) identifying and managing withdrawal symptoms patients may experience.
  Interventions: Behavioral: Computer-Assisted Preoperative CBT Intervention (PAINTrainer)
- Treatment-as-usual (control) (No Intervention): Patients scheduled to undergo total joint arthroplasty at the study site are automatically enrolled in a mandatory 4-hour education class delivered by a nurse educator or physical therapist. Utilizing an in-person Powerpoint presentation format, patients are informed about pre-habilitation exercises to do prior to surgery; what to expect the day of surgery; the multimodal analgesia protocol used in the perioperative period; options for anesthesia and analgesia; and the expectation of physical therapy after surgery.

INTERVENTIONS:
Behavioral: Computer-Assisted Preoperative CBT Intervention (PAINTrainer) — Subjects will be asked to complete eight (8) 30- to 45-minute educational sessions during the 4 weeks prior to your surgery. In addition to the computer based training sessions, there is a motivational interviewing component that requires subjects to meet with a member of the study team weekly for a total of four (4) 30- to 45-minute meetings to help manage opioid medication use. It is expected that subject participation in this arm of the study will be a total of 12 hours over the course of the entire study.
  Arms: Computer-Assisted Preoperative CBT Intervention

SUMMARY:
A significant number of patients develop chronic post-surgical pain (CPSP) following knee replacement surgery. Proposed is the testing of a novel computer-assisted behavioral intervention integrating motivational interviewing in the 4 weeks prior to surgery to address the risk factors for CPSP, with the expectation that severity of post-op pain and the incidence of CPSP will be reduced.

DETAILED DESCRIPTION:
A significant number of patients develop chronic post-surgical pain following knee joint replacement surgery, and the risk factors for this problematic outcome have been identified. Proposed is the development and preliminary efficacy testing of a novel computer-assisted cognitive behavioral intervention integrating motivational interviewing delivered in the four weeks prior to surgery to address these risk factors, with the expectation that both the severity of post-operative pain and the subsequent incidence of chronic post-surgical pain will be reduced. In that chronic post-surgical pain brings with it diminished functionality and quality of life, ongoing opioid use, and direct patient costs, it is critical that interventions aimed at mitigating its development are implemented and evaluated in the clinical setting.

In a sample of adults over the age of 21 with chronic pain undergoing a planned TKA, the objectives of this randomized clinical trial are to:

1. Add a motivational interviewing component to a validated computer-assisted CBT intervention for chronic pain (painTRAINER) to encourage opioid tapering, if applicable, and program adherence in the 4 weeks prior to surgery in patients scheduled to undergo a TKA.
2. Describe the efficacy of the 4-week targeted pre-operative CBT intervention in 45 TKA patients to decrease preoperative chronic pain severity, preoperative opioid consumption, and symptoms of depression, anxiety and pain catastrophizing prior to surgery in comparison to 45 TKA patients randomized to treatment-as-usual.
3. Describe the effects of a 4-week targeted pre-operative CBT intervention in 45 TKA patients on 48hr post-operative pain severity, and 3- and 6-month rates of CPSP in comparison to 45 TKA patients randomized to treatment-as-usual.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age > 21 years
2. Chronic non-malignant pain of at least 3 months duration
3. Morphine equivalent daily dose (MEDD) > 40 milligrams for at least 3 months
4. Able to enroll at least 4 weeks prior to planned surgery
5. Able to speak, read and comprehend in English at the 6th grade or higher proficiency

Exclusion Criteria:

1. Pain of malignant origin
2. Current or past history of opioid use disorder (including those on medication-assisted therapy)
3. Revision of TKA
4. Comorbid CNS disease such as dementia, HIV, psychosis, poorly controlled bipolar disorder or any condition interfering with informed consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin D Cheatle, PhD, Principal Investigator — University of Pennsylvania; Peggy Compton, RN, PhD, FAAN, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Penn Medicine University City, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Penn Medicine Radnor, Radnor, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
All records will be kept strictly confidential. No one except the researchers will know the subjects are in a research study. Data forms for the collection of health and study data will be coded with each subject's unique identification number. No data form will identify the participants by name. Hardcopies of data forms will be kept in locked files with keys held only by the study investigators. All electronic data will be stored with the password and firewall protected REDCap data collection and management system of the U Penn School of Nursing. No presentation or publication of the results of this study will refer to the individual participants or present information that would identify any participant. All persons working on the proposed work will have completed HIPAA training and the Collaborative Institutional Training Initiative (CITI) Basic Courses in the Protection of Human Research Subjects and Biomedical Focus Responsible Conduct of Research (RCR) modules.

REFERENCES:
- [Background] Inacio MCS, Paxton EW, Graves SE, Namba RS, Nemes S. Projected increase in total knee arthroplasty in the United States - an alternative projection model. Osteoarthritis Cartilage. 2017 Nov;25(11):1797-1803. doi: 10.1016/j.joca.2017.07.022. Epub 2017 Aug 8. PMID 28801208
- [Background] Sloan M, Premkumar A, Sheth NP. Projected Volume of Primary Total Joint Arthroplasty in the U.S., 2014 to 2030. J Bone Joint Surg Am. 2018 Sep 5;100(17):1455-1460. doi: 10.2106/JBJS.17.01617. PMID 30180053
- [Background] Lewis GN, Rice DA, McNair PJ, Kluger M. Predictors of persistent pain after total knee arthroplasty: a systematic review and meta-analysis. Br J Anaesth. 2015 Apr;114(4):551-61. doi: 10.1093/bja/aeu441. Epub 2014 Dec 26. PMID 25542191
- [Background] Petersen KK, Simonsen O, Laursen MB, Nielsen TA, Rasmussen S, Arendt-Nielsen L. Chronic postoperative pain after primary and revision total knee arthroplasty. Clin J Pain. 2015 Jan;31(1):1-6. doi: 10.1097/AJP.0000000000000146. PMID 25485953
- [Background] Petersen KK, Graven-Nielsen T, Simonsen O, Laursen MB, Arendt-Nielsen L. Preoperative pain mechanisms assessed by cuff algometry are associated with chronic postoperative pain relief after total knee replacement. Pain. 2016 Jul;157(7):1400-1406. doi: 10.1097/j.pain.0000000000000531. PMID 27331347
- [Background] Schug SA, Bruce J. Risk stratification for the development of chronic postsurgical pain. Pain Rep. 2017 Oct 31;2(6):e627. doi: 10.1097/PR9.0000000000000627. eCollection 2017 Nov. PMID 29392241
- [Background] Lavand'homme P. Transition from acute to chronic pain after surgery. Pain. 2017 Apr;158 Suppl 1:S50-S54. doi: 10.1097/j.pain.0000000000000809. No abstract available. PMID 28134653
- [Background] Richebe P, Capdevila X, Rivat C. Persistent Postsurgical Pain: Pathophysiology and Preventative Pharmacologic Considerations. Anesthesiology. 2018 Sep;129(3):590-607. doi: 10.1097/ALN.0000000000002238. PMID 29738328
- [Background] Goesling J, Moser SE, Zaidi B, Hassett AL, Hilliard P, Hallstrom B, Clauw DJ, Brummett CM. Trends and predictors of opioid use after total knee and total hip arthroplasty. Pain. 2016 Jun;157(6):1259-1265. doi: 10.1097/j.pain.0000000000000516. PMID 26871536
- [Background] Westermann RW, Anthony CA, Bedard N, Glass N, Bollier M, Hettrich CM, Wolf BR. Opioid Consumption After Rotator Cuff Repair. Arthroscopy. 2017 Aug;33(8):1467-1472. doi: 10.1016/j.arthro.2017.03.016. Epub 2017 May 29. PMID 28571723
- [Background] Parsons B, Schaefer C, Mann R, Sadosky A, Daniel S, Nalamachu S, Stacey BR, Nieshoff EC, Tuchman M, Anschel A. Economic and humanistic burden of post-trauma and post-surgical neuropathic pain among adults in the United States. J Pain Res. 2013 Jun 17;6:459-69. doi: 10.2147/JPR.S44939. Print 2013. PMID 23825931
- [Background] Katz J, Seltzer Z. Transition from acute to chronic postsurgical pain: risk factors and protective factors. Expert Rev Neurother. 2009 May;9(5):723-44. doi: 10.1586/ern.09.20. PMID 19402781
- [Background] Borsook D, Youssef AM, Simons L, Elman I, Eccleston C. When pain gets stuck: the evolution of pain chronification and treatment resistance. Pain. 2018 Dec;159(12):2421-2436. doi: 10.1097/j.pain.0000000000001401. PMID 30234696
- [Background] Althaus A, Hinrichs-Rocker A, Chapman R, Arranz Becker O, Lefering R, Simanski C, Weber F, Moser KH, Joppich R, Trojan S, Gutzeit N, Neugebauer E. Development of a risk index for the prediction of chronic post-surgical pain. Eur J Pain. 2012 Jul;16(6):901-10. doi: 10.1002/j.1532-2149.2011.00090.x. Epub 2011 Dec 23. PMID 22337572
- [Background] Buvanendran A, Della Valle CJ, Kroin JS, Shah M, Moric M, Tuman KJ, McCarthy RJ. Acute postoperative pain is an independent predictor of chronic postsurgical pain following total knee arthroplasty at 6 months: a prospective cohort study. Reg Anesth Pain Med. 2019 Mar;44(3):e100036. doi: 10.1136/rapm-2018-100036. Epub 2019 Feb 15. PMID 30770420
- [Background] Eisenach JC, Brennan TJ. Pain after surgery. Pain. 2018 Jun;159(6):1010-1011. doi: 10.1097/j.pain.0000000000001223. No abstract available. PMID 29768304
- [Background] Raja SN, Jensen TS. Predicting postoperative pain based on preoperative pain perception: are we doing better than the weatherman? Anesthesiology. 2010 Jun;112(6):1311-2. doi: 10.1097/ALN.0b013e3181dcd5cc. No abstract available. PMID 20502114
- [Background] McDonald S, Page MJ, Beringer K, Wasiak J, Sprowson A. Preoperative education for hip or knee replacement. Cochrane Database Syst Rev. 2014 May 13;2014(5):CD003526. doi: 10.1002/14651858.CD003526.pub3. PMID 24820247
- [Background] Riddle DL, Keefe FJ, Ang DC, Slover J, Jensen MP, Bair MJ, Kroenke K, Perera RA, Reed SD, McKee D, Dumenci L. Pain Coping Skills Training for Patients Who Catastrophize About Pain Prior to Knee Arthroplasty: A Multisite Randomized Clinical Trial. J Bone Joint Surg Am. 2019 Feb 6;101(3):218-227. doi: 10.2106/JBJS.18.00621. PMID 30730481
- [Background] Gibson E, Sabo MT. Can pain catastrophizing be changed in surgical patients? A scoping review. Can J Surg. 2018 Oct 1;61(5):311-318. doi: 10.1503/cjs.015417. PMID 30246983
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain - United States, 2016. MMWR Recomm Rep. 2016 Mar 18;65(1):1-49. doi: 10.15585/mmwr.rr6501e1. PMID 26987082
- [Background] Schug SA, Lavand'homme P, Barke A, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic postsurgical or posttraumatic pain. Pain. 2019 Jan;160(1):45-52. doi: 10.1097/j.pain.0000000000001413. PMID 30586070
- [Background] Borsook D, Kussman BD, George E, Becerra LR, Burke DW. Surgically induced neuropathic pain: understanding the perioperative process. Ann Surg. 2013 Mar;257(3):403-12. doi: 10.1097/SLA.0b013e3182701a7b. PMID 23059501
- [Background] Suzan E, Pud D, Eisenberg E. A crucial administration timing separates between beneficial and counterproductive effects of opioids on postoperative pain. Pain. 2018 Aug;159(8):1438-1440. doi: 10.1097/j.pain.0000000000001200. No abstract available. PMID 29521812
- [Background] McAnally H. Rationale for and approach to preoperative opioid weaning: a preoperative optimization protocol. Perioper Med (Lond). 2017 Nov 22;6:19. doi: 10.1186/s13741-017-0079-y. eCollection 2017. PMID 29201359
- [Background] Glare P, Aubrey KR, Myles PS. Transition from acute to chronic pain after surgery. Lancet. 2019 Apr 13;393(10180):1537-1546. doi: 10.1016/S0140-6736(19)30352-6. PMID 30983589
- [Background] Weber L, Yeomans DC, Tzabazis A. Opioid-induced hyperalgesia in clinical anesthesia practice: what has remained from theoretical concepts and experimental studies? Curr Opin Anaesthesiol. 2017 Aug;30(4):458-465. doi: 10.1097/ACO.0000000000000485. PMID 28590258
- [Background] Beck JS. Cognitive behavior therapy: Basics and beyond (2nd ed.). (2011) New York, NY: The Guilford Press.
- [Background] Turk DC, Flor H. Etiological theories and treatments for chronic back pain. II. Psychological models and interventions. Pain. 1984 Jul;19(3):209-233. doi: 10.1016/0304-3959(84)90001-0. PMID 6236417
- [Background] Knoerl R, Lavoie Smith EM, Weisberg J. Chronic Pain and Cognitive Behavioral Therapy: An Integrative Review. West J Nurs Res. 2016 May;38(5):596-628. doi: 10.1177/0193945915615869. Epub 2015 Nov 24. PMID 26604219
- [Background] Baez S, Hoch MC, Hoch JM. Evaluation of Cognitive Behavioral Interventions and Psychoeducation Implemented by Rehabilitation Specialists to Treat Fear-Avoidance Beliefs in Patients With Low Back Pain: A Systematic Review. Arch Phys Med Rehabil. 2018 Nov;99(11):2287-2298. doi: 10.1016/j.apmr.2017.11.003. Epub 2017 Dec 14. PMID 29247627
- [Background] Vugts MAP, Joosen MCW, van der Geer JE, Zedlitz AMEE, Vrijhoef HJM. The effectiveness of various computer-based interventions for patients with chronic pain or functional somatic syndromes: A systematic review and meta-analysis. PLoS One. 2018 May 16;13(5):e0196467. doi: 10.1371/journal.pone.0196467. eCollection 2018. PMID 29768436
- [Background] Eccleston C, Hearn L, Williams AC. Psychological therapies for the management of chronic neuropathic pain in adults. Cochrane Database Syst Rev. 2015 Oct 29;2015(10):CD011259. doi: 10.1002/14651858.CD011259.pub2. PMID 26513427
- [Background] Macea DD, Gajos K, Daglia Calil YA, Fregni F. The efficacy of Web-based cognitive behavioral interventions for chronic pain: a systematic review and meta-analysis. J Pain. 2010 Oct;11(10):917-29. doi: 10.1016/j.jpain.2010.06.005. Epub 2010 Jul 22. PMID 20650691
- [Background] Bender JL, Radhakrishnan A, Diorio C, Englesakis M, Jadad AR. Can pain be managed through the Internet? A systematic review of randomized controlled trials. Pain. 2011 Aug;152(8):1740-1750. doi: 10.1016/j.pain.2011.02.012. Epub 2011 May 11. PMID 21565446
- [Background] Aggarwal VR, Fu Y, Main CJ, Wu J. The effectiveness of self-management interventions in adults with chronic orofacial pain: A systematic review, meta-analysis and meta-regression. Eur J Pain. 2019 May;23(5):849-865. doi: 10.1002/ejp.1358. Epub 2019 Feb 7. PMID 30620145
- [Background] Monticone M, Ambrosini E, Cedraschi C, Rocca B, Fiorentini R, Restelli M, Gianola S, Ferrante S, Zanoli G, Moja L. Cognitive-behavioral Treatment for Subacute and Chronic Neck Pain: A Cochrane Review. Spine (Phila Pa 1976). 2015 Oct 1;40(19):1495-504. doi: 10.1097/BRS.0000000000001052. PMID 26192729
- [Background] Ehde DM, Dillworth TM, Turner JA. Cognitive-behavioral therapy for individuals with chronic pain: efficacy, innovations, and directions for research. Am Psychol. 2014 Feb-Mar;69(2):153-66. doi: 10.1037/a0035747. PMID 24547801
- [Background] Rini C, Porter LS, Somers TJ, McKee DC, DeVellis RF, Smith M, Winkel G, Ahern DK, Goldman R, Stiller JL, Mariani C, Patterson C, Jordan JM, Caldwell DS, Keefe FJ. Automated Internet-based pain coping skills training to manage osteoarthritis pain: a randomized controlled trial. Pain. 2015 May;156(5):837-848. doi: 10.1097/j.pain.0000000000000121. PMID 25734997
- [Background] Bennell KL, Nelligan R, Dobson F, Rini C, Keefe F, Kasza J, French S, Bryant C, Dalwood A, Abbott JH, Hinman RS. Effectiveness of an Internet-Delivered Exercise and Pain-Coping Skills Training Intervention for Persons With Chronic Knee Pain: A Randomized Trial. Ann Intern Med. 2017 Apr 4;166(7):453-462. doi: 10.7326/M16-1714. Epub 2017 Feb 21. PMID 28241215
- [Background] Bennell KL, Nelligan RK, Rini C, Keefe FJ, Kasza J, French S, Forbes A, Dobson F, Abbott JH, Dalwood A, Harris A, Vicenzino B, Hodges PW, Hinman RS. Effects of internet-based pain coping skills training before home exercise for individuals with hip osteoarthritis (HOPE trial): a randomised controlled trial. Pain. 2018 Sep;159(9):1833-1842. doi: 10.1097/j.pain.0000000000001281. PMID 29794609
- [Background] Cassin SE, Sockalingam S, Du C, Wnuk S, Hawa R, Parikh SV. A pilot randomized controlled trial of telephone-based cognitive behavioural therapy for preoperative bariatric surgery patients. Behav Res Ther. 2016 May;80:17-22. doi: 10.1016/j.brat.2016.03.001. Epub 2016 Mar 10. PMID 26990279
- [Background] Gade H, Friborg O, Rosenvinge JH, Smastuen MC, Hjelmesaeth J. The Impact of a Preoperative Cognitive Behavioural Therapy (CBT) on Dysfunctional Eating Behaviours, Affective Symptoms and Body Weight 1 Year after Bariatric Surgery: A Randomised Controlled Trial. Obes Surg. 2015 Nov;25(11):2112-9. doi: 10.1007/s11695-015-1673-z. PMID 25893651
- [Background] Lotzke H, Brisby H, Gutke A, Hagg O, Jakobsson M, Smeets R, Lundberg M. A Person-Centered Prehabilitation Program Based on Cognitive-Behavioral Physical Therapy for Patients Scheduled for Lumbar Fusion Surgery: A Randomized Controlled Trial. Phys Ther. 2019 Aug 1;99(8):1069-1088. doi: 10.1093/ptj/pzz020. PMID 30951604
- [Background] Wang L, Lee M, Zhang Z, Moodie J, Cheng D, Martin J. Does preoperative rehabilitation for patients planning to undergo joint replacement surgery improve outcomes? A systematic review and meta-analysis of randomised controlled trials. BMJ Open. 2016 Feb 2;6(2):e009857. doi: 10.1136/bmjopen-2015-009857. PMID 26839013
- [Background] das Nair R, Mhizha-Murira JR, Anderson P, Carpenter H, Clarke S, Groves S, Leighton P, Scammell BE, Topcu G, Walsh DA, Lincoln NB. Home-based pre-surgical psychological intervention for knee osteoarthritis (HAPPiKNEES): a feasibility randomized controlled trial. Clin Rehabil. 2018 Jun;32(6):777-789. doi: 10.1177/0269215518755426. Epub 2018 Feb 9. PMID 29424236
- [Background] Eccleston C, Fisher E, Thomas KH, Hearn L, Derry S, Stannard C, Knaggs R, Moore RA. Interventions for the reduction of prescribed opioid use in chronic non-cancer pain. Cochrane Database Syst Rev. 2017 Nov 13;11(11):CD010323. doi: 10.1002/14651858.CD010323.pub3. PMID 29130474
- [Background] Jung HJ, Yu ES, Kim JH. Combined Program of Cognitive-Behavioral Therapy for Insomnia and Medication Tapering in Cancer Patients: A Clinic-Based Pilot Study. Behav Sleep Med. 2020 May-Jun;18(3):386-395. doi: 10.1080/15402002.2019.1597718. Epub 2019 Apr 9. PMID 30966825
- [Background] Butler SF, Budman SH, Fernandez KC, Houle B, Benoit C, Katz N, Jamison RN. Development and validation of the Current Opioid Misuse Measure. Pain. 2007 Jul;130(1-2):144-56. doi: 10.1016/j.pain.2007.01.014. Epub 2007 May 9. PMID 17493754
- [Background] Cleeland CS. Measurement of pain by subjective report. In: Chapman CR, Loeser JD, editors. Issues in Pain Measurement. New York: Raven Press; pp. 391-403, 1989 Advances in Pain Research and Therapy; Vol. 12.
- [Background] Sullivan MJ, Bishop SR, Pivik J. The Pain Catastrophizing Scale: Development and Validation. Psychological Assessment 1995; 7(4): 524-532.
- [Background] Littell RC, Milli GA, Stroup WW, Wolfinger RD. SAS System for Mixed Models, Cary, NC: SAS Institute Inc., 1996, pp. 633.
- [Background] SAS Institute Inc. 2013. Base SAS® 9.4 Procedures Guide: Statistical Procedures, Second Edition. Cary, NC: SAS Institute Inc
- [Background] Little RJA. Modeling the drop-out mechanism in repeated-measures studies. Journal of the American Statistical Association. 1995;90:1112-21.
- [Background] Allison PD. Missing Data. Sage University Papers Series on Quantitative Applications in the Social Sciences, 2001; 07-136. Thousand Oaks, CA: Sage.
- See also: Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030 — https://www.ncbi.nlm.nih.gov/pubmed/17403800
- See also: Health Measures Website — http://www.healthmeasures.net/explore-measurement-systems/promis
- See also: Opioid Taper Decision Tool — https://www.pbm.va.gov/AcademicDetailingService/Documents/Pain_Opioid_Taper_Tool_IB_10_939_P96820.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Started | 27 | 27
Completed | 20 | 20
Not Completed | 7 | 7
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (7.69) | 57 (8.33) | 56 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Opioid morphine equivalents/day [Mean (Standard Deviation); unit: Opioid morphine equivalents/day] | 15.8 (36.36) | 11.4 (24.98) | 13.6 (30.87)

OUTCOME MEASURES:

1. Primary Outcome: Preoperative Chronic Pain Severity
Description: The severity of preoperative chronic pain will be evaluated with the Brief Pain Inventory (BPI), along two dimensions: intensity and interference. Pain intensity is rated on a 0 (no pain) to 10 (worst pain imaginable) scale as the worst in the past 24 hours, least in the past 24 hours, average pain and current pain. Pain interference is measured in 7 areas: general activity, mood, walking ability, work, sleep, enjoyment of life and relationships on a 0 (no interference) to 10 (interferes completely) scale. The composite mean of these scores are used as a pain interference score. BPI scores will be collected at baseline and compared to those collected just prior to surgery and at 3- and 6-month follow-up. Higher composite mean scores represent more pain interference (worse outcome).
Time Frame: prior to surgery, approximately 6 weeks following baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Number analyzed (Participants) | 20 | 20
units on a scale | 4.6 (2.13) | 4.4 (2.31)

2. Secondary Outcome: Preoperative Opioid Use
Description: Preoperative opioid use, if applicable, will be measured by converting to morphine equivalent daily dose (MEDD) at baseline and prior to surgery if the patients are still taking opioids.
Time Frame: prior to surgery, approximately 6 weeks following baseline
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Number analyzed (Participants) | 20 | 20
mg | 15.8 (36.36) | 11.4 (24.98)

3. Secondary Outcome: Post-operative Opioid Use
Description: Post-operative opioid use will be measured, if applicable, by converting to morphine equivalent daily dose (MEDD) at 48 hours post-operatively and 3- and 6-months follow up if the patients are still taking opioids.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Number analyzed (Participants) | 20 | 20
mg | 11.4 (31.58) | 12.0 (29.60)

4. Secondary Outcome: Pre-Op Depression
Description: To measure symptoms of depression, PROMIS® (Patient-Reported Outcomes Measurement Information System) depression person-centered scale will be utilized at baseline and pre-operation. Scores range from 8 to 40 with higher scores indicating greater severity of depression (worse outcome).
Time Frame: pre-operation, approximately 6 weeks following baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Number analyzed (Participants) | 20 | 20
score on a scale | 10.6 (3.69) | 11.2 (4.69)

5. Secondary Outcome: Post-Op Depression
Description: To measure symptoms of depression, the PROMIS® (Patient-Reported Outcomes Measurement Information System) depression person-centered scale will be utilized at 3- and 6-months post-operation. Scores range from 8 to 40 with higher scores indicating greater severity of depression (worse outcome).
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Number analyzed (Participants) | 20 | 20
score on a scale | 8.5 (1.02) | 10.6 (4.60)

6. Secondary Outcome: Pre-Op Anxiety
Description: To measure symptoms of anxiety, the PROMIS® (Patient-Reported Outcomes Measurement Information System) anxiety person-centered scale will be utilized at baseline and pre-operation. Scores range from 8 to 40, with higher scores indicating more severe anxiety (worse outcome).
Time Frame: pre-operation, approximately 6 weeks following baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Number analyzed (Participants) | 20 | 20
score on a scale | 13.0 (6.78) | 12.4 (5.27)

7. Secondary Outcome: Post-Op Anxiety
Description: To measure symptoms of anxiety, the PROMIS® (Patient-Reported Outcomes Measurement Information System) anxiety person-centered scale will be utilized at 3 and 6 months post-operation. Scores range from 8 to 40, with higher scores indicating more severe anxiety (worse outcome).
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Number analyzed (Participants) | 20 | 20
score on a scale | 9.1 (3.66) | 10.8 (7.12)

8. Secondary Outcome: Pre-Op Catastrophizing
Description: Pain catastrophizing will be measured by the Pain Catastrophizing Scale (PCS). The PCS is a 13-item self-report scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time). Scale scores range from 0 to 52; higher scores represent more pain catastrophizing (worse outcome).
Time Frame: pre-operation, approximately 6 weeks following baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Number analyzed (Participants) | 20 | 20
score on a scale | 10.8 (7.90) | 12.2 (11.17)

9. Secondary Outcome: Post-Op Pain Severity
Description: Severity of post-operative pain will be operationalized as responses on a visual analogue pain scale (VAS). The VAS ranges from 0 (no pain) to 10 (worst pain imaginable), and pain scores are collected every 4 hours as part of routine practice. These will be averaged over the first 48 hours post-operatively. Higher scores represent more severe post-operative pain (worse outcome).
Time Frame: 48 hours post-operatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Number analyzed (Participants) | 20 | 20
units on a scale | 4.6 (2.18) | 4.8 (1.98)

10. Secondary Outcome: Chronic Post-Surgical Pain
Description: To evaluate for the presence of chronic post-surgical pain (CPSP), subjects will be asked at 3- and 6-months if they have pain in the surgical site that developed or increased in intensity following the surgery utilizing a checklist based upon the IASP definition of CPSP (Appendix). This is a dichotomous measure with respondents reporting whether pain is absent (0) or present (1). A response of 1 (present) indicates that pain is present (a worse outcome).
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Number analyzed (Participants) | 20 | 20
Participants | 6 | 4

11. Secondary Outcome: Post-operative Chronic Pain Intensity
Description: Pain intensity is rated on a 0 (no pain) to 10 (worst pain imaginable) scale as the average pain intensity in the past 24 hours. Higher scores represent more severe pain (worse outcome).
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
Number analyzed (Participants) | 20 | 20
units on a scale | 3.1 (1.90) | 3.7 (2.59)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Computer-Assisted Preoperative CBT Intervention | Treatment-as-usual (Control)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT04814992/Prot_SAP_000.pdf